CLINICAL TRIAL: NCT00042575
Title: Protocol F1J-US-HMBY Dose Escalation, Double-Blind Treatment With Duloxetine Hydrochloride Once Daily Dosing for Evaluation of Safety in Major Depression
Brief Title: Dose Escalation, Double-Blind Treatment With Duloxetine Hydrochloride Once Daily Dosing for Evaluation of Safety in Major Depression
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 6475; F1J-US-HMBY
Record Dates: First submitted 2002-07-31; First posted 2002-08-05 (Estimated); Last update posted 2006-07-19 (Estimated); Status verified 2006-07

CONDITIONS: Major Depressive Disorder
Keywords: Sad, blue, lack of energy, depressed, hopelessness, guilt
MeSH Terms: conditions — Depressive Disorder, Major; Fatigue; Consciousness Disorders | interventions — Duloxetine Hydrochloride

INTERVENTIONS:
Drug: Duloxetine

SUMMARY:
The Purposes of this Study are to determine:

The safety of duloxetine and any side effects that might be associated with it.

Whether duloxetine can help patients with major depression.

It is possible that information collected during this study will be analyzed by the sponsor in the future to evaluate duloxetine for other possible uses or for other medical or scientific purposes other than those currently proposed.

Duloxetine might not have any good effects for you.

ELIGIBILITY:
Inclusion Criteria:

* You must be at least 18 years old.
* You must be diagnosed with major depressive disorder
* You must be able to visit the doctor's office once a week to once every 2 weeks for a total of 8 weeks.

Exclusion Criteria:

* You are a woman and are pregnant or breastfeeding.
* You have a current or previous major psychiatric disorder other than depression, such as bipolar disorder, schizophrenia, or other psychotic disorder.
* You have a history of alcohol or drug dependence or abuse within the past 6 months.
* You are allergic to the study drug or you have experienced allergic reactions when taking several medications at once.
* You have a serious medical illness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120
Dates: Start 2002-06; Study Completion 2002-08

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - Trumbull, Connecticut
  - Lafayette, Indiana
  - Gaithersburg, Maryland
  - Belmont, Massachusetts
  - Omaha, Nebraska
  - Albuquerque, New Mexico
  - Staten Island, New York
  - Salt Lake City, Utah
  - Bellevue, Washington

REFERENCES:
- [Derived] Wohlreich MM, Mallinckrodt CH, Prakash A, Watkin JG, Carter WP. Duloxetine for the treatment of major depressive disorder: safety and tolerability associated with dose escalation. Depress Anxiety. 2007;24(1):41-52. doi: 10.1002/da.20209. PMID 16845641